CLINICAL TRIAL: NCT04044638
Title: Eight Week Strength Training Reduces Blood Pressure of Middle Age Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Regional do Cariri (Other)
Responsible Party: Principal Investigator, Alfredo Anderson Teixeira de Araujo, Master of Science, Universidade Regional do Cariri
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2.821.574
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Blood Pressure; Resistance Training; Women

STUDY DESIGN:
Intervention Model Description: The sample consisted of 14 women, which were divided into two groups: young group (YG = 7) and middle age group (MAG = 7).
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Young Group (Experimental): Young women who underwent 8 weeks of training and had their blood pressure checked at baseline and after 4 and 8 weeks of training.
  Resistance training sessions were held 3 times a week, in which each session lasted 60 minutes and was performed for a period of 8 weeks. Each session consisted of 10-minute warm-up, shortly after, starting the exercises in the form of alternating circuit by segment, as: machine bench press, extension chair, high pull (front), flexor table, direct curl, leg press, triceps pulley, adductor, abdominal, abductor and calf. In all 10 exercises, 3 sets of 8 to 12 repetitions were performed, with an interval of 60 seconds between sets and intensity of 12 arbitrary units (a.u.) to 14 a.u., measured by the rate perception effort scale.
  Interventions: Other: Resistance trainining
- Middle-aged Group (Experimental): Middle-aged women women who underwent 8 weeks of training and had their blood pressure checked at baseline and after 4 and 8 weeks of training.
  Resistance training sessions were held 3 times a week, in which each session lasted 60 minutes and was performed for a period of 8 weeks. Each session consisted of 10-minute warm-up, shortly after, starting the exercises in the form of alternating circuit by segment, as: machine bench press, extension chair, high pull (front), flexor table, direct curl, leg press, triceps pulley, adductor, abdominal, abductor and calf. In all 10 exercises, 3 sets of 8 to 12 repetitions were performed, with an interval of 60 seconds between sets and intensity of 12 arbitrary units (a.u.) to 14 a.u., measured by the rate perception effort scale.
  Interventions: Other: Resistance trainining

INTERVENTIONS:
Other: Resistance trainining — Resistance training sessions were held 3 times a week, in which each session lasted 60 minutes and was performed for a period of 8 weeks. Each session consisted of 10-minute warm-up, shortly after, starting the exercises in the form of alternating circuit by segment, as: machine bench press, extension chair, high pull (front), flexor table, direct curl, leg press, triceps pulley, adductor, abdominal, abductor and calf. In all 10 exercises, 3 sets of 8 to 12 repetitions were performed, with an interval of 60 seconds between sets and intensity of 12 arbitrary units (a.u.) to 14 a.u., measured by the rate perception effort scale. In the first, fourth and eighth week, pre-exercise blood pressure (BP) was verified, in which the participants sat for a period of 10 minutes at rest, in a comfortable chair, with legs uncrossed, feet flat on the floor, back leaning on the chair, left arm at heart level and palm up to measure BP using a G * Tech-branded automatic digital device (MASTER model).

SUMMARY:
Introduction: Strength training (ST) is an important non-pharmacological means to reduce blood pressure (BP). Objective: To verify the pressure response of women after 8 weeks of ST. Method: Fourteen women were divided into young group (YG) and middle age (MAG) and submitted to ST for 8 weeks, lasting 60 minutes in 11 alternating exercises per segment with intensity of 12 to 13 on the subjective perception scale of effort. BP was verified at weeks 1, 4 and 8.

DETAILED DESCRIPTION:
The sample consisted of 14 women, which were divided into two groups: young group (YG = 7) and middle age group (MAG = 7). Inclusion criteria were: females aged 18 to 59 years, sedentary or who had not been engaged in any physical activity in the last 6 months, and the availability of time three times a week in the afternoon shift. Exclusion criteria were: morbid obesity (BMI> 40 kg.m-2), presenting any osteo-articular dysfunction.

After the adaptation period, resistance exercise sessions were started, which were performed 3 times a week on alternate days, in which each session lasted 60 minutes, and performed for a period of 8 weeks. Each session consisted of 10-minute warm-up on the treadmill or bicycle, shortly after, starting the exercises in the form of alternating circuit by segment, as: machine bench press, extension chair, high pull (front), flexor table, direct curl, leg press, triceps pulley, adductor, abdominal, abductor and calf. In all 10 exercises, 3 sets of 8 to 12 repetitions were performed, with an interval of 60 seconds between sets and intensity of 12 arbitrary units (a.u.) to 14 a.u., measured by the rate perception effort scale. In the first, fourth and eighth week, pre-exercise blood pressure (BP) was verified, in which the participants sat for a period of 10 minutes at rest, in a comfortable chair, with legs uncrossed, feet flat on the floor, back leaning on the chair, left arm at heart level and palm up1 to measure BP using a G * Tech-branded automatic digital device (MASTER MA100 model).

ELIGIBILITY:
Inclusion Criteria:

* Females between 18 and 59 years old, sedentary or who had not been engaged in any physical activity in the last 6 months, plus the availability of time three times a week in the afternoon shift.

Exclusion Criteria:

* Morbid obesity (BMI> 40 kg.m-2), presenting any osteo-articular dysfunction that limited the performance of exercises in strength training, women who were classified in category 3 (known serious disease) after risk stratification of the College American of Sports Medicine and also, who presented cardiovascular diseases, autonomic neuropathy, diabetes and hypertension controlled or not.

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2018-04-02 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Blood pressure | Four weeks
  Increased blood pressure in young group and reduced blood pressure in middle age group
Blood pressure | Eight weeks
  Increased blood pressure in young group and reduced blood pressure in middle age group

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Anderson T de Araujo, MSc, Principal Investigator — Universidade Regional do Cariri
Locations (1):
- Alfredo Anderson Teixeira de Araujo, Juazeiro do Norte, Ceará, Brazil

IPD SHARING:
Plan to Share IPD: No